CLINICAL TRIAL: NCT03703583
Title: Infant Feeding Practice and Gut Comfort: a Multi-country, Cross-sectional Observational Study
Brief Title: Infant Feeding Practice and Gut Comfort Study
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 17.12.INF
Record Dates: First submitted 2018-10-04; First posted 2018-10-12 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Healthy Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exclusively/predominantly Breastfeeding group
  Interventions: Other: There is no intervention in this observational study.
- Exclusively/predominantly Formula feeding group
  Interventions: Other: There is no intervention in this observational study.

INTERVENTIONS:
Other: There is no intervention in this observational study. — There is no intervention in this observational study.

SUMMARY:
Multi-country, cross-sectional, observational study in diverse geographic locations all over the world.

DETAILED DESCRIPTION:
This is a cross-sectional single time point study. Infants and caregivers who come to a clinic for a routine health visit who wish to participate in the study by signing the consent form and meet all inclusion criteria/exclusion criteria will be enrolled.

At the visit, a research staff member will assist the parents to complete (i) Feeding Practice and Gut Comfort Questionnaire and (ii) Infant Gastrointestinal Symptom (IGSQ)-13 items. Additionally, infant's anthropometrics (weight, length, head circumference) will be recorded. These anthropometrics will be measured by the researcher as part of the routine visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full term (37-42 weeks of gestation) singleton infant.
* Postnatal age ≥ 6 weeks and ≤ 4 months
* Parent as primary Caregiver and ≥ 18 years old
* Exclusively/predominantly breastfeeding or exclusively/predominantly formula feeding of the same type/brand, for at least the past 2 weeks.
* Evidence of personally signed and dated informed consent document by the infant's parent(s).

Exclusion Criteria:

* Chronic illness necessitating medical follow up
* Acute ongoing or recent (last 2 weeks) illness necessitating medical follow up
* Any known case of food allergy (e.g milk)
* Caregivers who are not likely to comply with the study procedures

Ages: 6 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy normal developing male and female full-term infants
Sampling Method: Non-Probability Sample
Enrollment: 2804 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
An index score of overall GI symptom burden | single time point between 6 weeks to 4 months
  Measured by Validated, standardized infant Gastrointestinal Symptom Questionnaire (IGSQ-13)

SECONDARY OUTCOMES:
GI Symptoms | single time point between 6 weeks to 4 months
  measured by IGSQ-13 questionnaires (An overall index score is calculated from 13 questions in the questionnaire as a measure of total GI symptom burden. The values for the IGSQ index score can range from 13 (low GI burden) to 65 (high GI burden))
Stool characteristics | one day recall before study visit
  measured by Feeding Practice and Gut Comfort Questionnaire (frequency and consistency)
Physician-reported and parent-reported Colic | Single time point between 6 weeks to 4 months
  measured by Feeding Practice and Gut Comfort Questionnaire based on ROME IV diagnosis criteria. Effect of feeding group on the prevalence of colic will be assessed by logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Vandenplas, Study Chair — Universitair Ziekenhuis Brussel
Locations (16):
- Egypt (6):
  - Alexandria University, Alexandria
  - Assuit University, Asyut
  - Ain Shams University, Cairo
  - Cairo University, Cairo
  - Tanta University, Tanta
  - Zagazig University, Zagazig
- India (3):
  - Apollo Children's Hospital, Chennai
  - ICH Hospital, Kolkata
  - Dr Praveen Gokhales Childrens Clinic and Vaccination Centre, Thane
- Faculty of Medicine Universitas Gadjah Mada, Yogyakarta, Indonesia
- University of Malaya, Kuala Lumpur, Malaysia
- Pakistan (4):
  - PIMS, Islamabad
  - National Institute of Child Health, Karachi
  - The Children Hospital & Institute of Child Health, Lahore
  - BBH, Rawalpindi
- St.Luke'S College of Medicine, Quezon City, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Happy Tummy Consortium; Lavalle L, Sauvageot N, Cercamondi CI, Egli D, Jankovic I, Vandenplas Y. Infant feeding practice and gastrointestinal tolerance: a real-world, multi-country, cross-sectional observational study. BMC Pediatr. 2022 Dec 14;22(1):714. doi: 10.1186/s12887-022-03763-8. PMID 36514058